CLINICAL TRIAL: NCT05173662
Title: The Effect of Pain Management Education on The Mothers on The Use of Nonpharmacological Practices and Anxiety Level in Heel Stick in Newborn
Brief Title: The Effect of Pain Management Education on The Mothers in Newborn
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Fatma Taş Arslan, Professor, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SelcukU-11-2021
Record Dates: First submitted 2021-11-29; First posted 2021-12-30 (Actual); Last update posted 2021-12-30 (Actual); Status verified 2021-12

CONDITIONS: Pain; Procedural Pain; Infant ALL
Keywords: pain; procedural; newborn; heel blood collection procedure; Education on nonpharmacological methods
MeSH Terms: conditions — Pain; Pain, Procedural

STUDY DESIGN:
Intervention Model Description: Intervention Group Education was given about non-pharmacological methods that can be applied during the heel blood collection procedure in newborns and a brochure was given.
  Control group: no intervention was made.
Who Masked: Outcomes Assessor
Masking Description: In order to avoid bias in the evaluation of the data, the analysis of the coded data in terms of groups was done by an independent statistician. After the statistical analyzes were completed and the research report was written, the researcher explained the coding of the intervention and control groups. In this way, single blindness was achieved.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): To the mothers in this group; At least 12 hours before the heel blood collection (guthrie screening test), training was given, lasting 25 minutes, on average, through the training brochure on non-pharmacological pain management prepared by the researcher. The training was carried out in a language that the mother could understand, in the form of direct lectures and questions and answers, using the visuals in the brochure. In the training content; There are five non-pharmacological methods. These;
  * Expressed breast milk
  * Wrapping
  * Skin-to-skin contact
  * Cuddling
  * They are methods of making calming sounds.
  Interventions: Procedure: Providing education and brochures on non-pharmacological methods that can be applied during the heel blood collection process
- Control Group (No Intervention): In the control group, as in the clinical routine, the heel stick procedure was performed in the newborn's own bed next to his mother. No other action has been applied.

INTERVENTIONS:
Procedure: Providing education and brochures on non-pharmacological methods that can be applied during the heel blood collection process — Theeduvation initiative was implemented by the researcher at least 12 hours ago in the mothers' room and a brochure was given about the education.
  Arms: Intervention Group

SUMMARY:
The aim of this study was to determine the effect of non-pharmacological pain management education given to mothers on the use of non-pharmacological methods and anxiety levels of mothers during routine heel blood collection (guthrie screening test) in term newborns.

H0= There was no difference between the intervention group who received non-pharmacological pain management education and the control group's level of anxiety and use of non-pharmacological applications.

H1= The use of non-pharmacological methods is different between the intervention group and the control group that received non-pharmacological pain management education.

H2= Anxiety scores of the intervention group that received non-pharmacological pain management education and the control group were different.

H3= Some characteristics and anxiety levels of mothers have an effect on their use of non-pharmacological methods.

It was carried out between July - September 2021 at the Akşehir State Hospital Gynecology and Obstetrics Clinic, which serves in the Akşehir district of Konya province.

DETAILED DESCRIPTION:
In this study was to determine the effect of pain management education on mothers' use of non-pharmacological methods and anxiety levels during newborn heel blood screening.

This study was designed as parallel group, pre-test and post-test randomized controlled trial.

Based on 80% power and 95% confidence level, the sample size was calculated as 32 infants for each group, a total of 64 infants (G*Power 3.1.9.2).

Randomization In this study, stratified randomization method was applied. Eight blocks of four were created with the permutation-blocked randomization method.

With the computer program (randomized.org), the numbers from 1 to 6 were listed 8 times (6,3,5,2,2,6,6,5) and the combinations were sorted according to this group, and assignments were made to the intervention and control groups.

Blinding The researcher and participant (mothers) could not be blinded since the researcher had to provide training and manage the process before the application. In order to avoid bias in the evaluation of the data, the analysis of the coded data in terms of groups was done by an independent statistician. After the statistical analyzes were completed and the research report was written, the researcher explained the coding of the intervention and control groups. In this way, single blindness was achieved.

In the collection of research data; Introductory Information Form, Non-pharmacological Method Application Checklist and Spielberger State Anxiety Inventory were used. In addition, the mothers in the intervention group were given a brochure on Nonpharmacological Pain Management Education Nonpharmacological Pain Management Education Brochure

This brochure was prepared by the researcher in line with the literature .The brochure contains methods for non-pharmacological pain management that can be applied during procedural painful interventions in newborns. These methods are; expressed breast milk, hugging, skin-to-skin contact, cuddling, calming sounds. The brochure contains information and drawings about the methods. The drawings were created by Architect Merve Özkald. Opinions were received from five experts in terms of the content, language, design and visual suitability of the brochure and the Content Validity Index (CGI) was calculated as 0.890.

Data collection Voluntary Informing Consent Form was obtained from the mothers before the study, and the Introductory Information Form was collected from the mothers by the researcher by face-to-face interview method. Between the dates of the study, mothers of newborns who met the inclusion criteria were randomly assigned to intervention and control groups. Heel blood collection in all newborns; The study was carried out between the 24th and 48th hours of the baby's life, in the gynecology and obstetrics clinic, only in the room where the mother and baby stay together, without any intervention to the baby, by removing the clothes from the lower part of the baby in its natural position.

The heel blood collection procedure was applied in such a way that the baby was next to the mother. No non-pharmacological method was used in routine practice during the procedure.

In this study; The heel blood collection procedure was performed by the same nurse working in the NICU for each infant at one time and by taking the same amount of blood from each infant on average.

At least half an hour before the heel blood collection, it was ensured that the babies were fed and their diapers were clean. During the blood collection process; Standardization of the blood collection technique used, the area where the blood was taken (outer side of the right heel), the needle used in the procedure (needle number 21), environmental factors (such as heat, light, noise), used antiseptic solution (70% alcohol) provided.

To the mothers in the intervention group; At least 12 hours before the heel blood collection (guthrie screening test), information was given by the researcher (FU) about the purpose of the heel blood collection procedure and the application process, and the questions, if any, were answered. Afterwards, an average of 25 minutes of education was given through the training brochure prepared by the researcher on non-pharmacological pain management. The education was carried out in a language that the mother could understand, in the form of direct lectures and questions and answers, using the visuals in the brochure.

The mothers in the control group, on the other hand, were informed by the researcher about the purpose of the heel blood collection procedure and the application process at least 12 hours before the guthrie screening test, and their questions were answered, if any, and no other application was made.

ELIGIBILITY:
Inclusion Criteria:

For newborns;

* Being a healthy term newborn (born at 38-42 weeks of gestation)
* A blood sample will be taken for the Guthrie screening test.
* Having the mother with the baby (Gynecology and Obstetrics Clinic) for mothers;
* Volunteering to participate in the study
* Ability to read and write Turkish
* Being over 18 years old

Exclusion Criteria:

For newborns;

* Having a congenital anomaly
* Having received any analgesia before the procedure
* IInability to draw blood in one go for mothers;
* Rejection of heel blood collection voluntarily
* Existence of any obstacle that may make communication difficult

Ages: 38 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2021-07-10 (Actual); Primary Completion 2021-09-24 (Actual); Study Completion 2021-11-24 (Actual)

PRIMARY OUTCOMES:
The mothers' use of non-pharmacological methods | After the process first 10 minute
  The mothers' use of non-pharmacological methods during heel blood collection. These methods are; expressed breast milk, hugging, skin-to-skin contact, cuddling, calming sounds. The cases of using the methods were determined as yes and no for each method.

SECONDARY OUTCOMES:
State anxiety level scores of mothers | Pre-test 5-10 minutes before the process and 10 minutes after the process
  The State and Trait Anxiety Inventory (STAI) was developed by Spielberger in 1983.
  The STAI consists of two subscales of 20 questions about state and trait anxiety.
  All questions are in a four-point Likert type. The scores of both subscales are summed separately and a total score between 20 and 80 is obtained.
  Higher scores indicate a higher level of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Fulya Unvar, Study Chair — Konya Aksehir State Hospital
Locations (2):
- Turkey (Türkiye) (2):
  - Selcuk University, Konya, Selcuklu
  - Selcuk University, Konya

REFERENCES:
- [Derived] Unvar F, Tas Arslan F. Effectiveness of maternal-targeted training on nonpharmacologic pain management on heel stick sampling: A randomized controlled trial. J Pediatr Nurs. 2023 Nov-Dec;73:e477-e483. doi: 10.1016/j.pedn.2023.10.018. Epub 2023 Nov 3. PMID 37923615